CLINICAL TRIAL: NCT03875820
Title: FRAME: A Phase I Trial of the Combination of Defactinib (VS-6063) (FAK Inhibitor) and VS-6766 (RO5126766) (CH5126776) (a Dual RAF/MEK Inhibitor) in Patients With Advanced Solid Tumours
Brief Title: Phase I Trial of Defactinib and VS-6766.
Acronym: FRAME
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Institute of Cancer Research, United Kingdom (Other)
Collaborators: Verastem, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CCR4642; 2017-001035-39 (EudraCT Number)
Record Dates: First submitted 2018-11-15; First posted 2019-03-15 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: NSCLC; Low Grade Serous Ovarian Cancer; Endometrioid Carcinoma; Pancreatic Cancer
Keywords: KRAS G12V; RAS; RAF
MeSH Terms: conditions — Carcinoma, Endometrioid; Pancreatic Neoplasms | interventions — RO5126766; defactinib

STUDY DESIGN:
Intervention Model Description: The dose escalation phase will enrol patients with advanced RAS mutant solid tumours.
  In the dose expansion phase, patients are assigned to one of the following cohorts based on their diagnosis:
  * KRAS mutant NSCLC cohort
  * LGSOC cohort
  * RAS mutant CRC cohort
  * Advanced RAS mutant solid tumour cohort - patients in this cohort must have biopsiable disease, be willing and consent to undergo biopsies at three time-points.
  * KRAS G12V mutant NSCLC cohort
  * RAS/RAF mutant endometrioid cohort
  * Pancreatic cohort
Masking Description: Non-randomised: Participants are expressly assigned by phase of study and diagnosis.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Dose Escalation Phase (Experimental): Escalating doses of VS-6766 (RO5126766) and Defactinib (VS-6063) were evaluated in patients with advanced solid tumours to establish the recommended phase II dose. Dose escalation followed a 3+3 design with a maximum of four patient cohorts.
  This arm is now complete.
  Interventions: Drug: VS-6766; Drug: Defactinib
- Dose Expansion KRAS mutant NSCLC Cohort (Experimental): The dose expansion phase will evaluate the recommended phase II dose of the combination of VS-6766 (RO5126766) and Defactinib (VS-6063), as decided in the dose escalation phase in patients with KRAS mutant NSCLC (20 patients).
  This arm is now complete.
  Interventions: Drug: VS-6766; Drug: Defactinib
- Dose Expansion biopsy cohort (Experimental): The dose expansion phase will evaluate the recommended phase II dose of the combination of VS-6766 (RO5126766) and Defactinib (VS-6063), as decided in the dose escalation phase in patients advanced RAS mutant solid tumours with biopsiable disease (6 patients).
  This arm is now complete.
  Interventions: Drug: VS-6766; Drug: Defactinib
- Dose Expansion LGSOC cohort (Experimental): The dose expansion phase will evaluate the recommended phase II dose of the combination of VS-6766 (RO5126766) and Defactinib (VS-6063), as decided in the dose escalation phase in patients with LGSOC (20 patients).
  Interventions: Drug: VS-6766; Drug: Defactinib
- Dose Expansion CRC cohort (Experimental): The dose expansion phase will evaluate the recommended phase II dose of the combination of VS-6766 (RO5126766) and Defactinib (VS-6063), as decided in the dose escalation phase in patients with CRC (10 patients).
  This arm is now complete.
  Interventions: Drug: VS-6766; Drug: Defactinib
- Dose Expansion KRAS G12V mutant NSCLC cohort (Experimental): The dose expansion phase will evaluate the recommended phase II dose of the combination of VS-6766 (RO5126766) and Defactinib (VS-6063), as decided in the dose escalation phase in patients with KRAS G12V mutant NSCLC (10 patients).
  Interventions: Drug: VS-6766; Drug: Defactinib
- Dose Expansion RAS/RAF mutant endometrioid cancer cohort (Experimental): The dose expansion phase will evaluate the recommended phase II dose of the combination of VS-6766 (RO5126766) and Defactinib (VS-6063), as decided in the dose escalation phase in patients with RAS/RAF mutant endometrioid subtype of gynaecological cancers (ovarian, endometrial, endometriosis-related) (10 patients).
  Interventions: Drug: VS-6766; Drug: Defactinib
- Dose Expansion pancreatic cancer (Experimental): The dose expansion phase will evaluate the recommended phase II dose of the combination of VS-6766 (RO5126766) and Defactinib (VS-6063), as decided in the dose escalation phase in patients with pancreatic cancer (10 patients).
  Interventions: Drug: VS-6766; Drug: Defactinib

INTERVENTIONS:
Drug: VS-6766 — VS-6766 will be supplied as 0.8mg hypromellose (HPMC) capsules for oral administration. The capsule fill consists of VS-6766 and the inactive ingredients mannitol and magnesium stearate.
  VS-6766 will be administered on a twice weekly (Monday and Thursday or Tuesday and Friday) schedule for 3 weeks followed by 1 week off in every 4 week cycle, under fasting conditions (approximately 1 hour prior or 2 hours after a meal). The starting dose, based on the previous Phase I trial will be 3.2 mg given orally as a single daily dose. This can be escalated to a maximum of 4mg (as per dose escalation rules in the protocol).
  Other Names: RO5126766; CH5126766
Drug: Defactinib — Defactinib is formulated as a white to off-white oval tablet for oral administration and supplied in single unit dose strength of 200 mg in 120 cc (HDPE) bottles. In addition to Defactinib, formulation components include microcrystalline cellulose, lactose monohydrate, sodium starch glycolate, and magnesium stearate.
  Patients will receive Defactinib orally immediately after a meal twice daily (approximately every 12 hours) for 3 weeks followed by 1 week off in every 4 week cycle. The starting dose will be 200mg. This can be escalated to a maximum of 400mg (as per dose escalation rules in the protocol).
  Other Names: VS-6063

SUMMARY:
This is a multi-centre, investigator-initiated, dose escalation, Phase I trial of the combination of the FAK inhibitor, Defactinib (VS-6063), and the dual RAF/MEK inhibitor, VS-6766 (RO5126766) in patients with advanced solid tumours. VS-6766 (RO5126766) is the same compound as CH5126766.

There are two parts to this study, the dose escalation phase and the dose expansion phase. In the dose escalation phase, cohorts of 3 to 6 patients will be enrolled to determine the maximum tolerated dose (MTD) and recommended Phase II dose (RP2D). This will be followed by a dose expansion phase to further characterise the safety and tolerability and to assess the pharmacodynamic activity of the combination.

DETAILED DESCRIPTION:
This is a multi-centre, investigator-initiated, dose escalation, Phase I trial of the combination of the FAK inhibitor, Defactinib, and the dual RAF/MEK inhibitor, VS-6766 in patients with advanced solid tumours.

There are two parts to this study, the dose escalation phase and the dose expansion phase. In the dose escalation phase, cohorts of 3 to 6 patients were enrolled to determine the maximum tolerated dose (MTD) and recommended Phase II dose (RP2D). Up to 24 patients with solid tumours were treated in the dose escalation phase of this study.

The dose escalation phase is now closed to recruitment.

This will be followed by a dose expansion phase of 86 patients to further characterise the safety and tolerability and to assess the pharmacodynamic activity of the combination.

The dose expansion phase is made up of 7 cohorts:

* 20 patients with KRAS mutant non-small-cell lung cancer (NSCLC);
* 7 patients with solid tumours (enriched for those with RAS mutations) willing to undergo biopsies at three time points throughout the study;
* 20 patients with low grade serous ovarian cancer (LGSOC);
* 10 patients with colorectal cancer (CRC);
* 10 patients with KRAS G12V mutant NSCLC;
* 10 patients with RAS/RAF mutant endometrioid subtype of gynaecological cancers (ovarian, endometrial, endometriosis related) and
* 10 patients with pancreatic cancer.

The following cohorts are still open to recruitment:

* Patients with low grade serous ovarian cancer (LGSOC);
* Patients with KRAS G12V mutant NSCLC;
* Patients with RAS/RAF mutant endometrioid subtype of gynaecological cancers (ovarian, endometrial, endometriosis-related) and
* Patients with pancreatic cancer.

Patients will take the two investigational medicinal products (IMPs) as follows:

VS-6766 will be administered orally twice a week on Monday/Thursday or Tuesday/Friday at least one hour prior or two hours after a meal. The starting dose of VS-6766 will be 3.2mg once a day, twice a week and can be escalated to a maximum of 4mg once a day, twice a week.

Defactinib will be administered orally twice a day immediately after a meal. The starting dose of Defactinib will be 200mg twice daily and can be escalated to a maximum of 400mg twice daily.

A cycle length is 4 weeks (28 days). Combination dosing (VS-6766 and Defactinib) will commence on Cycle 1 Day 1 for 3 weeks followed by one week without either drug in week 4 (i.e. 3 weeks on, 1 week off).

For patients consenting to optional biopsies, a run-in dose of VS-6766 will be administered on a single day anywhere between Days -7 to Day -3 in order to facilitate pharmacodynamic (PD) biomarker analysis. Therefore, for patients undergoing biopsies the first cycle will be 5 weeks long and subsequent cycles will consist of 4 weeks.

If this schedule is not tolerated, alternative schedules may be explored following discussion by the Safety Review Committee.

ELIGIBILITY:
Inclusion Criteria:

1. Dose escalation:

   Histologically or cytologically proven solid tumours, refractory to conventional treatment, or for which no conventional therapy exists or is declined by the patient enriching for patients with RAS mutant solid tumours.

   Dose expansion:

   Histologically or cytologically proven advanced non-small-cell lung cancer (NSCLC) with a documented KRAS mutation, refractory to conventional treatment, or for which no conventional therapy exists or is declined by the patient (20 patients).

   OR Histologically or cytologically proven advanced low grade serous ovarian cancer (LGSOC), refractory to conventional treatment, or for which no conventional therapy exists or is declined by the patient (20 patients).

   OR Histologically or cytologically proven advanced colorectal cancer (CRC) with a documented RAS mutation, refractory to conventional treatment, or for which no conventional therapy exists or is declined by the patient (10 patients).

   OR Histologically or cytologically proven RAS mutant solid tumours, refractory to conventional treatment, or for which no conventional therapy exists or is declined by the patient. Patient must have biopsiable disease, be willing and has consented to undergo biopsies at three time-points (6 patients).

   OR Histologically or cytologically proven advanced pancreatic cancer or metastatic pancreatic cancer, refractory to conventional treatment, or for which no conventional therapy exists or is declined by the patient (10 patients).

   OR Endometroid subtype of gynaecological cancers (ovarian, endometrial, endometriosis related) with a documented RAS or RAF mutation, refractory to conventional treatment, or for which no conventional therapy exists or is declined by the patient (10 patients).

   OR Histologically or cytologically proven advanced non-small-cell lung cancer (NSCLC) with a documented KRAS G12V specific mutation, refractory to conventional treatment, or for which no conventional therapy exists or is declined by the patient (10 patients).
2. Predicted life expectancy of at least 12 weeks
3. World Health Organisation (WHO) performance status of 0 or 1 (Appendix 1)
4. Haematological and biochemical indices within the ranges shown below. These measurements must be performed within one week (Day -7 to Day 1) before the patient goes in the trial.

   Haemoglobin (Hb) ≥ 9.0 g/dL Absolute neutrophil count (ANC) ≥ 1.5 x 109/L Platelet count ≥ 100 x 109/L Serum bilirubin ≤ 1.5 x upper limit of normal (ULN) Alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST)

   ≤ 2.5 x (ULN) unless raised due to tumour in which case up to 5 x ULN is permissible

   Either:

   Calculated creatinine clearance ≥ 50 mL/min (uncorrected value)

   Or:

   Serum creatinine ≤ 1.5 x ULN
5. Men and women aged 18 years or over.
6. Written (signed and dated) informed consent and be capable of co-operating with treatment and follow-up.
7. Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule.
8. Dose escalation: Measurable disease according to RECIST 1.1 or evaluable disease. All radiology studies must be performed within 28 days prior to registration.

   Dose expansion: Measurable disease according to RECIST 1.1, all radiology studies must be performed within 28 days prior to registration.
9. Corrected QT interval (QTc) < 470 ms (as calculated by the Fridericia correction formula, averaged over 3 ECGs).
10. Agrees to the use of archival paraffin embedded tissue and has archival tumour tissue available.

Exclusion Criteria:

1. Radiotherapy (except for palliative reasons), endocrine therapy, biological therapy, immunotherapy or chemotherapy during the previous four weeks (six weeks for nitrosoureas, Mitomycin-C) before treatment.
2. Ongoing toxic manifestations of previous treatments. Exceptions to this are alopecia or certain Grade 1 toxicities, which in the opinion of the Investigator and the DDU should not exclude the patient.
3. Known untreated or active central nervous system (CNS) metastases (progressing or requiring corticosteroids for symptomatic control). Patients with a history of treated CNS metastases are eligible, provided they meet all of the following criteria:

   * Evaluable or measurable disease outside the CNS is present.
   * Radiographic demonstration of improvement upon the completion of CNS-directed therapy and no evidence of interim progression between the completion of CNS-directed therapy and the baseline disease assessment for at least 28 days.
4. Ability to become pregnant (or already pregnant or lactating). However, those female patients who have a negative serum or urine pregnancy test before enrolment and agree to use two medically approved forms of contraception (oral, injected or implanted hormonal contraception and condom, have an intra-uterine device and condom, diaphragm with spermicidal gel and condom) from time of consent, during the trial and for six months afterwards are considered eligible.
5. Male patients with partners of child-bearing potential (unless they agree to take measures not to father children by using one form of medically approved contraception [condom plus spermicide] during the trial and for six months afterwards). Men with pregnant or lactating partners should be advised to use barrier method contraception (for example, condom plus spermicidal gel) to prevent exposure to the foetus or neonate.
6. Major surgery within 4 weeks prior to entry to the study (excluding placement of vascular access), or minor surgery within 2 weeks of entry into the study and from which the patient has not yet recovered.
7. Treatment with warfarin. Patients on warfarin for DVT/PE can be converted to LMWH.
8. Known history of Gilbert's Syndrome.
9. Acute or chronic pancreatitis.
10. At high medical risk because of non-malignant systemic disease including active uncontrolled infection.
11. Known to be serologically positive for hepatitis B, hepatitis C or human immunodeficiency virus (HIV).
12. Patients with the inability to swallow oral medications or impaired gastrointestinal absorption due to gastrectomy or active inflammatory bowel disease.
13. Concurrent ocular disorders:

    1. Patients with history of glaucoma, history of retinal vein occlusion (RVO), predisposing factors for RVO, including uncontrolled hypertension, uncontrolled diabetes
    2. Patient with history of retinal pathology or evidence of visible retinal pathology that is considered a risk factor for RVO, intraocular pressure > 21mm Hg as measured by tonometry, or other significant ocular pathology, such as anatomical abnormalities that increase the risk for RVO.
    3. Patients with a history of corneal erosion (instability of corneal epithelium), corneal degeneration, active or recurrent keratitis, and other forms of serious ocular surface inflammatory conditions.
14. Concurrent congestive heart failure, prior history of class III/ IV cardiac disease (New York Heart Association [NYHA] - refer to Appendix 4), myocardial infarction within the last 6 months, unstable arrhythmias, unstable angina or severe obstructive pulmonary disease.
15. Patients exposed to strong CYP3A4 and strong CYP2C9 inhibitors within 7 days prior to the first dose.

    N.B. Because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated list such as http://medicine.iupui.edu/clinpharm/ddis/table.aspx; medical reference texts such as the Physicians' Desk Reference may also provide this information.
16. Is a participant or plans to participate in another interventional clinical trial, whilst taking part in this Phase I study of VS-6766 in combination with Defactinib. Participation in an observational trial would be acceptable.
17. Symptoms of COVID-19 and/or documented current COVID-19 infection (the patient can be reassessed for eligibility following a full recovery and negative COVID-19 test).
18. Any other condition which in the Investigator's opinion would not make the patient a good candidate for the clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2017-12-12 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-10-31 (Estimated)

PRIMARY OUTCOMES:
To establish a dose for Phase II evaluation from the maximum tolerated dose of the combination of VS-6766 and Defactinib. | 12 months
  To determine the maximum dose at which no more than 1 of 6 patients at the same dose level experience a drug related toxicity (DLT) as specified in the protocol.
Measure Adverse Events according to CTCAE v4.0. | 6 months
  To assess the safety and toxicity profile of VS-6766 and Defactinib. To determine causality and grading severity of each adverse event by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.

SECONDARY OUTCOMES:
To characterise the pharmacokinetic profile of VS-6766 in combination with Defactinib. | 12 months
  Determination of the PK parameter Cmax of VS-6766 and Defactinib when dosed together.
To characterise the pharmacokinetic profile of VS-6766 in combination with Defactinib. | 12 months
  Determination of the PK parameter terminal half-life of VS-6766 and Defactinib when dosed together.
To characterise the pharmacokinetic profile of VS-6766 in combination with Defactinib. | 12 months
  Determination of the PK parameter area under the curve of VS-6766 and Defactinib when dosed together.

OTHER OUTCOMES:
To document any possible anti-tumour activity in patients. | 24 months
  Determination of disease response by RECIST criteria version 1.1 and collection of data related to progression free survival.
To study the pharmacodynamic profile of VS-6766 alone and in combination with Defactinib in pre-treatment and post-treatment biopsies and PBMCs. | 24 months
  Quantification of biomarkers such as p-MEK, p-ERK and p-FAK, E-cadherin and vimentin and enumeration of T cell populations which express CD8, CD4 and CD25.
To assess putative predictive biomarkers of response and resistance to the combination of VS-6766 and Defactinib. | 24 months
  Correlation of antitumour activity of the combination of VS-6766 and Defactinib with the detection of putative predictive biomarkers of response and resistance in archival tumours and plasma DNA.

CONTACTS AND LOCATIONS:
Overall Officials: Udai Banerji, FRCP, PhD, Principal Investigator — Institute of Cancer Research, United Kingdom
Locations (5):
- United Kingdom (5):
  - The Christie NHS Foundation Trust, Manchester, Greater Manchester
  - The Royal Marsden NHS Foundation Trust, Sutton, Surrey
  - The Royal Marsden NHS Foundation Trust - Gynecology Unit, London
  - The Newcastle Upon Tyne Hospitals NHS Foundation Trust - Freeman Hospital, Newcastle
  - The Royal Marsden NHS Foundation Trust - Gynecology Unit, Sutton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Banerjee S, Krebs MG, Greystoke A, Garces AI, Perez VS, Terbuch A, Shinde R, Caldwell R, Grochot R, Rouhifard M, Ruddle R, Gurel B, Swales K, Tunariu N, Prout T, Parmar M, Symeonides S, Rekowski J, Yap C, Sharp A, Paschalis A, Lopez J, Minchom A, de Bono JS, Banerji U. Defactinib with avutometinib in patients with solid tumors: the phase 1 FRAME trial. Nat Med. 2025 Sep;31(9):3074-3080. doi: 10.1038/s41591-025-03763-y. Epub 2025 Jun 27. PMID 40579546
- [Derived] Fard D, Giraudo E, Tamagnone L. Mind the (guidance) signals! Translational relevance of semaphorins, plexins, and neuropilins in pancreatic cancer. Trends Mol Med. 2023 Oct;29(10):817-829. doi: 10.1016/j.molmed.2023.07.009. Epub 2023 Aug 17. PMID 37598000